CLINICAL TRIAL: NCT06084871
Title: Patient Blood Management in Cardiac Surgery in Turkiye
Acronym: PaBMiCS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ERAS Turkey Association (Other)
Responsible Party: Sponsor
Other Study IDs: I11-657-22
Record Dates: First submitted 2023-10-10; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Coronary Artery Disease; Iron Deficiency Anemia
Keywords: Patient blood management; CABG; intravenous iron
MeSH Terms: conditions — Coronary Artery Disease; Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient Blood Management group: Three pillars of patient blood management will be applied
- Control group: Control

SUMMARY:
* Rationale and background: Surgical patients' transfusions have changed from replacing surgically lost blood with allogenic blood transfusions to implementing strategies that reduce transfusion requirements. Patient Blood Management (PBM) is designed to maintain hemoglobin concentration, optimize hemostasis, and minimize blood loss to improve patient outcomes. There is mounting evidence that multimodal PBM programs can improve postoperative outcomes and reduce perioperative blood transfusions and costs. The TULIP study in Turkey showed higher uses of blood transfusions in major surgical patients, including coronary artery surgeries in Turkey. The current studies also support the preoperative use of intravenous iron and/or vitamin B12/folic acid in major surgical patients. So, we aim to evaluate the efficacy of implantation of PBM in CABG surgeries in Turkey.
* Research question and objectives: Is it possible to decrease the amount of perioperative blood and blood products transfusions by implementing PBM in patients who underwent CABG surgeries? The primary objective of the study is to demonstrate the reduction in perioperative RBC units transfused, when PBM is implemented in cardiac surgery in Turkey. The secondary objectives are to evaluate the concurrent reduction of FFP, platelet and total blood products used as compared to a control group, length of hospital and ICU stay following the surgery.
* Study design: A prospective, multicenter, non-interventional study with a historical/retrospective control group.
* Population: Patients who are operated on for coronary artery bypass grafting.
* Variables: Demographic (age, sex), clinical (body mass index, comorbidities, ASA score, P-POSSUM score, Charlson Comorbidity Index), operative (type and duration of operations), laboratory (hemoglobin, platelet count, coagulation profile), laboratory for anemia (transferrin saturation, ferritin, creatinine clearance), preoperative treatment, transfusion data, and outcome (morbidity, mortality, lengths of hospital stay).
* Exposures: Preoperative IV iron treatment of anemia.
* Data sources: Medical data of the patients are obtained after entering a prespecified database (e-CRF) for the study subjects. For the control group, the medical data of the patients will be obtained retrospectively from the database of the TULIP study.
* Study size: Study group: A total of 368 patients from five different centers across Turkey. Control group: at least 368 patients from the same centers attending the TULIP study. Finally, 736 patients will be included for the study.

DETAILED DESCRIPTION:
Patient blood management (PBM) is defined as "the timely application of evidence-based medical and surgical concepts designed to maintain hemoglobin concentration, optimize haemostasis and minimize blood loss in an effort to improve patient's outcome" (1,2). Patient blood management has recently been introduced in several areas where blood transfusions are important, such as anaesthesiology, cardiac surgery, orthopedic surgery, or traumatology (3).

Its adoption has been recommended by the WHO since 2010, as well as by national health regulation agencies, international professional societies, and the European Commission (4-7). In literature, there is mounting evidence that multimodal PBM programs can be effective at improving postoperative outcomes and reducing perioperative blood transfusions and costs (8).

Turkish Society of Anaesthesiology and Reanimation (TARD) PBM Task Force has been working on this subject and studied transfusion practices in major surgery patients and the prevalence of perioperative anemia (9). In the TULIP study, unfortunately, high usage of transfusions in major surgical patients in Turkey was documented. As demonstrated in the TULIP study, one of the surgeries that had high transfusion use, was cardiac surgery. Speciﬁc procedures with the highest RBC use were also coronary artery bypass grafting (16.9% of all units). Low hemoglobin concentration was the most common indication for intra-operative RBC transfusion (57%).

Preoperative anemia is common in cardiac surgery, with a prevalence between 10% and 50% (depending on the applied definition). Using the standard World Health Organization definition, the prevalence of anemia in the adult cardiac surgery population seems to be around 20% to 30% (10). Preoperative anemia is an independent risk factor for the transfusion of RBC, postoperative morbidity, and mortality (11, 12). An analysis of 9,144 cardiac surgery patients demonstrated that patients with low hematocrit values (<25%) during surgery who were exposed to RBC transfusion had an increased morbidity (cardiac and renal) and hospital mortality (13). Preoperative anemia is mostly the result of inadequate erythropoiesis owing to iron deficiency, malnutrition, malabsorption, inflammation, bone marrow disorders, or chronic blood loss. Importantly, anemic patients with iron deficiency need to be identified as early as possible by the cardiologist, surgeon, or anesthesiologist. With the introduction of a special PBM anemia walk-in clinic, anemia management can be initiated at an early stage. This would allow for timely optimization of iron stores to compensate for iron deficiency (14) or other treatable forms of anemia. Diagnosis and treatment of preoperative anemia are currently not part of standard care but are a core element of PBM to increase Hb values in cardiac surgery patients. In recent years, many studies investigated preoperative anemia and its effects on the outcome of adult cardiac surgery patients (Table 1).

Table 1. Preoperative anemia and its effects on the outcome of adult cardiac surgery patients

Author Study Design Sample Size Primary Outcome

* Kulier et al. 2007 (14) Prospective, observational 5,065 Cardiac and noncardiac adverse events ↑
* van Straten et al. 2009 (15) Prospective, observational 10,025 Early and late mortality ↑
* Carrascal et al. 2010 (16) Cohort study (retrospective) 1,388 Red cell transfusion ↑ Hospital stay ↑
* Piednoir et al. 2011 (17) Cohort study (retrospective) 100 Transfusion rate ↑ Postoperative fatigue ↑
* Hung et al. 2011 (18) Cohort study (retrospective) 2,688 Transfusion ↑ Death ↑ ICU stay ↑
* David et al. 2013 (19) Cohort study (retrospective) 943 Transfusion rate ↑
* Kim et al. 2015 (20) Cohort study (retrospective) 712 Transfusion rates ↑ Morbidity ↑
* Hallward et al. 2016 (21) Cohort study (retrospective) 1,972 Blood transfusion ↑ ICU stay ↑ Hospital stay ↑

When the interventional studies investigating the effect of PBM in cardiac surgery patients are examined, the studies showing visible differences are shown in Table 2.

Table 2. The effect of PBM in cardiac surgery patients

Author Study Design Sample Size Intervention Primary Outcome

* Karkouti et al. 2006 (22) Randomized, interventional 31 Iron ± EPO Hb level →
* Cladellas et al. 2012 (23) Cohort study (retrospective) 134 EPO + IV iron Renal failure ↓ Red blood cell transfusion ↓
* Garrido-Martin et al. 2012 (24) Randomized, interventional 159 Oral or IV iron IV iron Hb level →
* Johansson et al. 2015 (25) Randomized, interventional 60 IV iron Hb level ↑
* Duce et al. 2017 (26) Cohort study retrospective 159 EPO vs. blood cell transfusion Mortality → Thrombotic events →
* Spahn et al. 2019 (27) Randomized, interventional 1,006 IV iron, erythropoietin alpha, vitamin B12 and folic acid Red blood cell transfusions ↓ Hb level ↑ Reticulocytes ↑ Reticulocyte Hb ↑

In literature, IV iron treatment is recommended for cardiac surgery patients. Examples of these studies can be given as follows: Iron supplementation, especially in combination with EPO is recommended when anemia of chronic disease is accompanied by iron deficiency with complete depletion of iron stores (28).

The Hb concentration after iron supplementation rise approximately 1 to 2 g/dL within 2 to 4 weeks. Very recently, a trial investigating the effect of ultra-short-term treatment (combination of iron, erythropoietin, vitamin B12, and folic acid administration) of 505 patients with iron deficiency or anemia undergoing cardiac surgery showed significantly reduced RBC transfusions, higher Hb concentration, higher reticulocyte count, and a higher reticulocytes Hb content during the first 7 days (27). This study suggests that an iron supplementation even immediately before cardiac surgery has beneficial effects, however, an early start to therapy could be more effective (29,30).

Whether different thresholds of Hb defining anemia in men and women lead to an undertreatment of female patients has been investigated in many studies and is the subject of current discussions. Most of these studies were conducted with cardiac surgery patients (31,32). The latest data show that women have worse outcomes compared with men having anemia.

Although other factors have an impact on this result (e.g., higher age, higher incidence of comorbidities, more acute and symptomatic stage in women), it is proposed that for all patients, regardless of sex, a Hb threshold of 13 g/dL should be applied (33). This is particularly important in those undergoing surgery with the use of cardiopulmonary bypass where dependent on the system, in most cases, the same volume of fluid is added to the pump. Perioperative bleeding has been shown to be an independent predictor of hospital mortality. In a study including more than 9000 patients undergoing cardiac surgery with CPB, massive blood loss (defined by the transfusion of at least five units of packed red blood cells on the day of surgery) was associated with an 8-fold increase in mortality (34). Other studies have also reported excess morbidity, particularly in terms of thromboembolic complications, infections, and higher rates of surgical re-exploration (35). Notably, surgical re-exploration and transfusion following bleeding are also associated with increased infection, mortality, and a longer stay in ICU and hospital (36,37).

Excessive postoperative hemorrhage in cardiac surgery has a significant economic impact: a retrospective German analysis of more than 1100 patients estimated its average additional cost to be €6251 per patient (38).

Oral iron therapy is inexpensive and easy to administer, but its gastrointestinal side effects limit the routine use of oral iron therapy (39). Several studies reported the good efficacy of intravenous iron therapy (IVIT) in increasing hemoglobin levels and reducing blood transfusions in patients with anemia (40-42). However, the recovery profiles according to the status of the disease or condition of the patients are controversial regarding the efficacy of IVIT in transfusion practices. While some elements of PBM have a strong evidence base in cardiac surgery, such as the use of tranexamic acid (TXA) and reduced transfusion thresholds (43,33), the evidence for preoperative anemia optimization with IVIT is less in Turkiye. Sert et al. from Turkiye, evaluated retrospectively the data of patients who underwent elective open-heart surgery. Their primary aim was to compare the patient outcomes, the requirement for transfusion, and the cost of transfusion between two different periods with and without PBM protocols. The authors found that the transfusion of unnecessary blood and blood products was reduced, and the cost decreased with the PBM protocol, although blood product usage did not affect 30-day mortality (44). It was observed that 37.1% of the patients were anemic, 50.6% were using anticoagulant drugs, and 78% had at least an additional disease. Although these factors were regarded as risk factors for transfusion, it was determined that patients with anemia had more frequently required transfusions than those without anemia.

In the general framework, five main risk factors for high risk of bleeding or transfusion are very consistently identified independently of the country: pre-operative anemia, prior cardiac surgery, clopidogrel 5 days or less before surgery, use of other P2Y12 inhibitors at any point, and thrombocytopenia <100.000 platelets/mm3. In conclusion, more efforts are needed to clarify and complement the currently available guidelines and to define a homogenous landscape for PBM practices implementation (45).

Potential barriers to the implementation of PBM are lack of knowledge, under-representation of anemia management in the education of young physicians, inadequate interpretation of controversial evidence, errors in reasoning, oversimplification, wide variations in belief, and lack of agreement of hospitals, self-efficiency, outcome expectancy, and stability of the previous practice (46).

Therefore, we plan to perform a large-scale, prospective study in which a well-designed PBM program is used to confirm the efficacy of perioperative IVIT in patients with CABG surgery. As a second step, PABMiCS study is proposed to identify the benefits of PBM implementation, including preoperative anemia management, in major cardiac surgeries in Turkiye.

ELIGIBILITY:
Inclusion Criteria:

* Signed patient informed consent
* Male or female patient 18-80 years old
* Patients scheduled for elective first time coronary artery bypass grafting (CABG)
* Antiplatelet treatment will be discontinued in patients on antiplatelet therapy and will be operated after wash-out time as recommended in the guidelines. If the patient needs to be operated before wash-out period completed, then the patient will be excluded from the study.
* Patients with confirmed iron deficiency anemia (IDA), defined as Hb 100-130 g/L, and serum ferritin < 100 ng/ml or TSAT < 20%.

Patients with iron deficiency anemia in the "PBM active group" will be taken into surgery 3 weeks after the treatment for study group.

Exclusion Criteria:

* Patients that undergo emergency surgical procedure
* Patients with non-iron deficiency anaemia (thalassemia, sickle cell anemia and etc)
* Patients with renal anemia (Hb < 130 g/L and CCL < 50 mL/min, irrespective of iron parameters) or any diagnosis that require EPO
* Patients with Hb < 100 g/L
* Patients with known anaphylactic/hypersensitivity reactions to parenteral iron products
* Patients with iron overload or disturbances in utilization of iron (e.g., haemochromatosis, hemosiderosis)
* Patients with ≥3 times increase in aspartate aminotransferase or alanine aminotransferase as per reference range
* Patients with excessive blood loss requiring massive transfusion (≥ 10 more red blood cell units)
* Patients with known myelodysplastic syndromes
* Patients with chronic kidney disease with an estimated CCL < 50 mL/min or with end-stage renal disease requiring scheduled dialysis
* Patients with known urinary tract infections with urea-splitting bacteria
* Any patient judged to lack the ability to give informed consent or perform the trial assessments (e.g., due to dementia)
* Women who are pregnant or breast feeding
* Intention to become pregnant during the course of the study
* Lack of safe contraception, defined as: Female participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases (Female participants who are surgically sterilized / hysterectomized or post-menopausal for longer than 2 years are not considered as being of child bearing potential),
* Known or suspected non-compliance, drug or alcohol abuse
* Patients who will be re-operated after being included in study
* Participation in another study with investigational drug within the 30 days preceding and during the present study.
* Patients receiving ≥10 units of RBCs within 24h from start of surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CABG with iron deficiency anemia
Sampling Method: Non-Probability Sample
Enrollment: 368 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Red blood cell transfusion | 7 days
  The reduction of perioperative RBC units transfused as a compared to a control group

SECONDARY OUTCOMES:
Length of ICU stay | 7 days
  The reduction of ICU stays as compared to a control group
Length of stay | 7 days
  The reduction of length of stay as compared to a control group

CONTACTS AND LOCATIONS:
Overall Officials: Onat Bermede, MD, Principal Investigator — Ankara University
Locations (1):
- Ankara University School of Medicine Heart Center, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided